CLINICAL TRIAL: NCT00570232
Title: Phase II Trial to Assess Target Oral Therapy as Adjuvant Chemoprevention in High-Risk Head and Neck Cancer
Brief Title: UAB 0718 - Phase II Trial to Assess Target Oral Therapy as Adjuvant Chemoprevention in High-Risk Head and Neck Cancer
Acronym: UAB0718
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Genentech, Inc. (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Eben Rosenthal, Professor of Surgery, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: F070824015; UAB 0718 (Other: UAB ComprehensiveCancerCenter ClinicalTrialsReviewCommittee)
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Head and Neck Cancer
Keywords: Resectable, recurrent head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tarceva (Other): All patients will be prescribed erlotinib 150mg daily
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — 150 mg per day by mouth for 12 months
  Other Names: Tarceva

SUMMARY:
The purpose of this study is to determine whether erlotinib will be effective in controlling cancer that has returned after treatment with salvage surgery and radiation. This study will also determine what effects, good and/or bad, this drug has on the participants.

DETAILED DESCRIPTION:
An investigator-initiated Phase II clinical trial of the safety and tolerability of erlotinib as an adjuvant therapy after definitive therapy via salvage surgery in head and neck cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed diagnosis of recurrent or second primary squamous cell carcinoma
2. Recurrence or second primary of the oral cavity, oropharynx, hypopharynx, or larynx. Recurrent neck metastasis with unknown primary is allowed
3. Prior radiation therapy for head and neck cancer
4. Disease must be considered surgically resectable or candidate for curative reirradiation
5. Adequate diagnostic workup
6. Zubrod Performance Status 0-2
7. Life expectancy 12 weeks
8. Age 19, 9. Adequate laboratory data.

Exclusion Criteria:

1. Prior invasive cancers other than head and neck cancer unless disease free for a minimum of 3 years. (Prior non-melanomatous skin cancer and previous carcinoma in situ are permissible)
2. Patients who are pregnant or lactating
3. Psychological condition that renders the patient unable to understand the informed consent
4. Any situation or condition that will interfere with adherence to study activities.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-12; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eben Rosenthal, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Tarceva: All patients will be prescribed Tarceva 150mg daily
  Erlotinib: 150 mg per day by mouth for 12 months
Period: Overall Study
Arm/Group | Tarceva
Started | 31
Completed | 8
Not Completed | 23
Not completed — Adverse Event | 10
Not completed — discontinued due to medical condition | 3
Not completed — discontinued due to recurrence | 8
Not completed — discontinued due to noncompliance | 2

BASELINE CHARACTERISTICS:
Arm/Group | Tarceva
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 18
ECOG performance status [Number; unit: participants] — ECOG PS 0 Fully active,able to carry on all predisease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory & able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory & capable of all selfcare but unable to carry out any work activities. Up & about more than 50% of waking hours
  3. Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair
  5. Dead The ECOG PS is in the public domain.
  participants
    0 | 18
    1 | 8
    2 | 2
    unknown | 3
Tumor Stage at Study Start - Primary Tumor Stage (T) [Number; unit: participants] — Classification of Malignant Tumors based on the American Joint Committee on Cancer (AJCC) staging criteria. T indicates tumor size, extent, or penetration (depth) of the tumor. T1 is the smallest/least advanced,while T4 is the largest/most advanced.
  participants
    T1 | 1
    T2 | 3
    T3 | 6
    T4 | 13
    not specified | 8
Tumor Stage at Study Start - Regional Metastasis (N) [Number; unit: participants] — Classification of Malignant Tumors based on the American Joint Committee on Cancer (AJCC) staging criteria. N indicates the number of lymph nodes with cancer or the location of the cancer-involved lymph nodes.
  N0 = no regional lymph node metastasis
  N1 = a single ipsilateral lymph node <3 cm in greatest dimension
  N2 = a single ipsilateral lymph nodes 3-6 cm in size OR multiple ipsilateral, bilateral, or contralateral lymph nodes <6 cm in greatest dimension
  N3 = a lymph node >6 cm in greatest dimension
  participants
    N0 | 18
    N1 | 2
    N2 | 2
    N3 | 1
    not specified | 8
Extent of recurrence [Number; unit: participants]
  Local | 21
  Regional | 5
  Locoregional | 5
Tumor subsite [Number; unit: participants] — location of primary tumor
  participants
    oral cavity | 11
    larynx | 7
    hypopharynx | 3
    oropharynx | 9
    unknown | 1
Procedure details [Number; unit: participants] — Number of participants who received coincident placement of tracheostomy or PEG tube during salvage surgery prior to enrollment
  participants
    Coincident tracheostomy | 13
    Coincident PEG | 11
    None | 7
Flap reconstruction [Number; unit: participants] — Number of participants who received flap reconstruction during salvage surgery prior to enrollment
  participants
    Yes | 27
    No | 4
Neck dissection [Number; unit: participants] — Number of participants who received a neck dissection (either unilateral or bilateral) during salvage surgery prior to enrollment
  participants
    Unilateral | 9
    Bilateral | 12
    None | 10
Histological tumor grade [Number; unit: participants]
  Well differentiated | 1
  Moderately differentiated | 14
  Poorly differentiated | 7
  Not specified | 9
Histological features [Number; unit: participants]
  Perineural invasion present | 10
  Lymphovascular invasion present | 4
  Positive lymph nodes | 4
  None | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Demonstrating the Safety and Tolerability of Long Term Erlotinib Treatment
Description: Number of participants who had the most frequently observed undesirable effects after exposure to study drug
Time Frame: 12 - 24 months
Measure: Number; unit: participants
Arm/Group | Tarceva
Number analyzed (Participants) | 31
participants
  rash | 26
  diarrhea | 22
  fatigue | 22
  nausea | 6
  vomiting | 6
  headache | 4

2. Primary Outcome: Percentage of Participants With Disease Free Status at 12 Months and 24 Months
Description: Percentage of participants who were disease free at 12 months (12 months after initiation of study drug treatment) and 24 months (12 months after completion of study drug treatment)
Time Frame: 12 - 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Tarceva
Number analyzed (Participants) | 31
percentage of participants
  disease free rate at 12 months | 54
  disease free rate at 24 months | 45

3. Secondary Outcome: Percentage of Participants Demonstrating Survival at 12 Months and 24 Months.
Description: Percentage of participants who were still alive at 12 months following completion of study drug therapy and at 24 months following completion of study drug therapy
Time Frame: 12 - 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Tarceva
Number analyzed (Participants) | 31
percentage of participants
  survival rate at 12 months | 61
  survival rate at 24 months | 56

ADVERSE EVENTS:
Arm/Group | Tarceva
Serious Adverse Events (participants affected / at risk) | 9/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tarceva (N=31)
pneumonia leading to respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pt hospitalized for respiratory failure and pneumonia felt releated to disease recurrence
bleeding from throat (Surgical and medical procedures) | 1 (1) — Pt hospitalized for throat bleeding felt related to disease progress
stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pt hospitalized for stridor and trach debulking, felt unrelated to study drug
Bell's Palsy (Nervous system disorders) | 1 (1) — Pt hospitalized and diagnosed with Bell's Palsy
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (2) — Pt hospitalized for pneumonia
cardiac stents placed (Cardiac disorders) | 1 (1) — Pt had cardiac stents placed; event deemed unrelated to protocol therapy
H pylori infection (Infections and infestations) | 1 (1) — Pt hospitalized for nausea and vomiting felt related to inadequate PEG and H pylori infection
myocardial infarction (Cardiac disorders) | 1 (1) — Pt hospitalized for MI felt possibly related to study drug
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pt hospitalized for septic shock and ARDS related to pneumonia; unrelated to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tarceva (N=31)
acniform rash (Skin and subcutaneous tissue disorders) | 26
fatigue (General disorders) | 22
diarrhea (Gastrointestinal disorders) | 22
hyperglycemia (Metabolism and nutrition disorders) | 21
anemia (Metabolism and nutrition disorders) | 13
dry skin (Skin and subcutaneous tissue disorders) | 12
hypoalbuminemia (Metabolism and nutrition disorders) | 7
nausea (Gastrointestinal disorders) | 6
vomiting (Gastrointestinal disorders) | 6
weight loss (Investigations) | 5
decreased platelet count (Metabolism and nutrition disorders) | 5
hyperkalemia (Metabolism and nutrition disorders) | 4
hypercalcemia (Metabolism and nutrition disorders) | 4
headache (Nervous system disorders) | 4
constipation (Gastrointestinal disorders) | 4
hyponatremia (Metabolism and nutrition disorders) | 4
hirsutism (Skin and subcutaneous tissue disorders) | 3
dyspepsia (Gastrointestinal disorders) | 3
depression (Psychiatric disorders) | 3
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
reflux (Gastrointestinal disorders) | 2
hypomagnesemia (Metabolism and nutrition disorders) | 2
alopecia (Skin and subcutaneous tissue disorders) | 2
hypophosphatemia (Metabolism and nutrition disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No